CLINICAL TRIAL: NCT00710736
Title: A Study of ARRY-334543 and Capecitabine in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-543-204
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — ARRY-334543; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARRY-334543 + capecitabine (Experimental)
  Interventions: Drug: ARRY-334543, EGFR/ErbB2 inhibitor; oral; Drug: Capecitabine, 5-fluorouracil prodrug; oral

INTERVENTIONS:
Drug: ARRY-334543, EGFR/ErbB2 inhibitor; oral — multiple dose, escalating
Drug: Capecitabine, 5-fluorouracil prodrug; oral — multiple dose, single schedule

SUMMARY:
This is a Phase 1 study during which patients with advanced/metastatic solid tumors will receive investigational study drug ARRY-334543 and capecitabine. Patients will receive increasing doses of study drug in combination with capecitabine in order to achieve the highest dose of study drug possible that will not cause unacceptable side effects. Patients will be followed to see what side effects the combination causes and what effectiveness the combination has, if any, in treating the cancer. Approximately 30 patients from the US and Canada will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of any advanced/metastatic cancer suitable for treatment with capecitabine. Pancreatic cancer is not allowed and patients with gastric or gastroesophageal junction (GEJ) cancer are only eligible if prior treatment did not include a total gastrectomy.
* Target lesions may be in a previously irradiated field only if progression of the lesion has been clearly documented.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2.
* Must be able to take and retain oral medications.
* Additional criteria exist.

Key Exclusion Criteria:

* Active concomitant malignancies.
* Uncontrolled or symptomatic brain metastases (if a patient has brain metastases and is on steroids, the steroid dose must be stable for at least 30 days).
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Requiring intravenous (IV) alimentation.
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C.
* Pregnancy or lactation.
* Chemotherapy, anticancer immunotherapy, monoclonal antibodies or biologics within 21 days prior to first dose of study drug.
* Anti-EGFR and/or ErbB2 small molecule targeted therapy or hormonal anticancer therapy within 14 days prior to first dose of study drug.
* History of any hypersensitivity to or intolerance of capecitabine or any of its components, or to fluorouracil or any fluoropyrimidine therapy.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of study drug in combination with capecitabine. | Duration of study
Characterize the safety profile of study drug in combination with capecitabine in terms of adverse events, clinical laboratory tests and electrocardiograms. | Duration of study
Characterize the pharmacokinetics (PK) of study drug and capecitabine. | Duration of study

SECONDARY OUTCOMES:
Assess the efficacy of the study drug in combination with capecitabine in terms of tumor response and changes in serological tumor markers. | Duration of study
Assess potential predictive biomarkers of clinical activity for the study drug in combination with capecitabine. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Roswell Park Cancer Institute, Buffalo, New York
- Canada (2):
  - British Columbia Cancer Agency- Centre for the Southern Interior, Kelowna, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario